CLINICAL TRIAL: NCT05545735
Title: Duration of Antibiotic Therapy for Early (DATE) Ventilator-Associated Pneumonia (VAP) Trial: A Surgical Infection Society Multicenter Randomized Clinical Trial of 4 vs. 7 Days of Definitive Antibiotic Therapy for Early VAP
Brief Title: The Duration of Antibiotic Therapy for Early (DATE) Ventilator Associated Pneumonia (VAP): 4 vs. 7 Days
Acronym: DATE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The rate of enrollment was slower than expected
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Jonathan Meizoso, Assistant Professor of Surgery, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20211211
Record Dates: First submitted 2022-09-12; First posted 2022-09-19 (Actual); Results first posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 4 Days of Antibiotics Group (Experimental): Participants will receive 4 days of antibiotic therapy administered as per the standard of care for the treatment of early ventilator associated pneumonia (VAP).
  Interventions: Drug: Standard of Care Antibiotic Therapy
- 7 Days of Antibiotics Group (Active Comparator): Participants will receive 7 days of antibiotic therapy administered as per the standard of care for the treatment of early ventilator associated pneumonia (VAP).
  Interventions: Drug: Standard of Care Antibiotic Therapy

INTERVENTIONS:
Drug: Standard of Care Antibiotic Therapy — Antibiotics will be administered as per the standard of care orally via tablet

SUMMARY:
The purpose of this study is to see if the amount of antibiotics given for ventilator-associated pneumonia (VAP) can be decreased in order to reduce the risk of adverse effects associated with antibiotics, while at the same time ensuring the participant's safety.

ELIGIBILITY:
Inclusion Criteria:

1. Surgical patient
2. Early VAP, defined as VAP occurring within 2 - 7 days of intubation (via endotracheal or tracheostomy tube) (9). VAP will be defined according to local institutional protocol.
3. Hospital length of stay (LOS) < 10 days at the time of VAP diagnosis.
4. Patients are willing to provide informed consent or their Legally Authorized Representative (LAR) is willing to provide informed consent on their behalf when the patient is unable (i.e., cognitively impaired from sedation on a ventilator)

Exclusion Criteria:

1. Age < 18 years
2. Prior episode of VAP for the index admission
3. VAP caused by any of the following pathogens:

   * Methicillin-resistant Staphylococcus aureus (MRSA)
   * Vancomycin-intermediate Staphylococcus aureus (VISA)
   * Pseudomonas aeruginosa
   * Vancomycin-resistant Enterococcus (VRE)
   * Acinetobacter baumanii
   * Stenotrophomonas maltophilia
   * Carbapenem-resistant Enterobacteriaceae (CRE)
   * Extended-spectrum beta lactamase-producing gram-negative bacilli
4. Causative pathogen not sensitive to choice of initial empiric antibiotic
5. Antibiotic therapy for > 5 of the last 10 days preceding VAP diagnosis
6. Septic shock, defined as evidence of tissue hypoperfusion after adequate volume expansion, due to infection, and requiring > 1 vasopressor (17)
7. Current or recent (within 30 days) use of immunosuppressive medications
8. LOS > 72 hours at a transferring facility
9. Pregnancy or lactation
10. Legal arrest or incarceration
11. Moribund state in which death is imminent
12. ECMO (Extracorporeal membrane oxygenation)
13. Extubation prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Meizoso, MD, MSPH, Principal Investigator — University of Miami
Locations (1):
- Jackson Memorial Hospital, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 4 Days of Antibiotics Group | 7 Days of Antibiotics Group
Started | 12 | 15
Completed | 12 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4 Days of Antibiotics Group | 7 Days of Antibiotics Group | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Continuous [Mean (Full Range); unit: years] | 51 [22 to 78] | 43 [19 to 71] | 47 [19 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 11 | 13 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 4 | 2 | 6
  Unknown or Not Reported | 3 | 6 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 7 | 11
Number of Subjects with causative pathogen sensitive to initial empiric antibiotic [Count of Participants; unit: Participants] | 12 | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Reoccurring VAP
Description: VAP recurrence will be reported as the number of participants with VAP occurring following completion of initial therapy.
Time Frame: Up to 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | 4 Days of Antibiotics Group | 7 Days of Antibiotics Group
Number analyzed (Participants) | 12 | 15
Participants | 5 | 7

2. Primary Outcome: Antibiotic Free Days
Description: The number of days where participant did not require the use of antibiotics
Time Frame: Up to 30 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 4 Days of Antibiotics Group | 7 Days of Antibiotics Group
Number analyzed (Participants) | 12 | 15
Days | 17.2 (7.7) | 14 (6.6)

3. Secondary Outcome: Number of Days of Antibiotic Exposure
Description: The number of days when the participant received antibiotics
Time Frame: Up to 30 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 4 Days of Antibiotics Group | 7 Days of Antibiotics Group
Number analyzed (Participants) | 12 | 15
Days | 12.8 (7.7) | 16 (6.6)

4. Secondary Outcome: Amount of Antibiotic Exposure
Description: Antibiotic exposure will be expressed as the total number of antibiotic days, defined as one antibiotic agent administered for one day. For example, if a patient receives two different antibiotics for five days, this equals 10 antibiotic days. The "number of antibiotics used" refers to the number of different antibiotic agents administered per day, not the number of individual doses or pills.
Time Frame: Up to 30 days
Measure: Mean (Standard Deviation); unit: Antibiotic Days
Arm/Group | 4 Days of Antibiotics Group | 7 Days of Antibiotics Group
Number analyzed (Participants) | 12 | 15
Antibiotic Days | 21.1 (13.4) | 23.8 (11.0)

5. Secondary Outcome: Clinical Improvement as Measured by the Change in Clinical Pulmonary Infection Score (CPIS) From the First Study Day to the Last
Description: Clinical improvement will be measured comparing the difference from the first study day to the last study day using daily Clinical Pulmonary Infection Score (CPIS) clinical score while enrolled in the study. CPIS has a total score ranging from 0 to 12 where a score of less than 6 indicates that the lung infection is considered controlled. A negative change may suggest improvement while a positive difference may suggest a worsening.
Time Frame: From baseline to the last study day, up to 30 days
Measure: Median (Full Range); unit: Change of score on a scale
Arm/Group | 4 Days of Antibiotics Group | 7 Days of Antibiotics Group
Number analyzed (Participants) | 12 | 15
Change of score on a scale | -2 [-4 to 3] | -1 [-7 to 1]

6. Secondary Outcome: Number of Participants With VAP Relapse
Description: VAP relapse will be reported as any recurrence of VAP caused by initial pathogen.
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 4 Days of Antibiotics Group | 7 Days of Antibiotics Group
Number analyzed (Participants) | 12 | 15
Participants | 1 | 4

7. Secondary Outcome: Ventilator-free Days
Description: The average number of days participants did not use a ventilator
Time Frame: Up to 30 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 4 Days of Antibiotics Group | 7 Days of Antibiotics Group
Number analyzed (Participants) | 12 | 15
Days | 17.7 (5.3) | 13.3 (11.1)

8. Secondary Outcome: The Number of Participants With Empyema
Description: The number of participants with empyema
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 4 Days of Antibiotics Group | 7 Days of Antibiotics Group
Number analyzed (Participants) | 12 | 15
Participants | 0 | 0

9. Secondary Outcome: The Number of Participants That Received a Tracheostomy
Description: The number of participants that received a tracheostomy
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 4 Days of Antibiotics Group | 7 Days of Antibiotics Group
Number analyzed (Participants) | 12 | 15
Participants | 2 | 8

10. Secondary Outcome: The Number of Participants With Non-pulmonary Infections
Description: The number of participants with Non-pulmonary infections
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | 4 Days of Antibiotics Group | 7 Days of Antibiotics Group
Number analyzed (Participants) | 12 | 15
Participants | 0 | 0

11. Secondary Outcome: ICU-free Days
Description: The average number of days participants were not in the ICU
Time Frame: Up to 30 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 4 Days of Antibiotics Group | 7 Days of Antibiotics Group
Number analyzed (Participants) | 12 | 15
Days | 11.8 (9.7) | 7.2 (6.4)

12. Secondary Outcome: Hospital Length Of Stay
Description: Number of days participant was admitted in the hospital
Time Frame: Up to 1 year
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 4 Days of Antibiotics Group | 7 Days of Antibiotics Group
Number analyzed (Participants) | 12 | 15
Days | 66.9 (108.1) | 33.7 (12.6)

13. Secondary Outcome: In-hospital Mortality
Description: The number of participants that died while admitted in the hospital will be reported
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | 4 Days of Antibiotics Group | 7 Days of Antibiotics Group
Number analyzed (Participants) | 12 | 15
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was assessed for up to 1 year. Serious and Other (Not Including Serious) Adverse Events were assessed for 30 days from admission or until hospital discharge, whichever occurred first.
Description: This patient population who require critical care support will experience a number of common aberrations in laboratory values, signs, and symptoms due to the severity of the underlying disease and the impact of standard therapies. These will not necessarily constitute an AE unless they require significant intervention, lead to discontinuation of study procedures, felt to be related to study procedures or are considered to be of concern in the Investigator's clinical judgment.
Arm/Group | 4 Days of Antibiotics Group | 7 Days of Antibiotics Group
All-Cause Mortality (participants affected / at risk) | 2/12 | 2/15
Serious Adverse Events (participants affected / at risk) | 2/12 | 5/15
Other Adverse Events (participants affected / at risk) | 0/12 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4 Days of Antibiotics Group (N=12) | 7 Days of Antibiotics Group (N=15)
Brain Death (Nervous system disorders) | 2 (2) | 2 (2) — Brain Death
Worsening Brain Bleed (Nervous system disorders) | 0 (0) | 1 (1) — Brain bleed became worse as compared to baseline
Above the Knee Amputation (Vascular disorders) | 0 (0) | 1 (1) — Amputation of the lower limb above the knee
Blood Stream Infection (Infections and infestations) | 0 (0) | 1 (1) — Blood Stream Infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT05545735/Prot_SAP_000.pdf